CLINICAL TRIAL: NCT05428332
Title: Examining the Efficacy of a Tri-Compartment Unloader Knee Brace During Physical Rehabilitation in Non-Surgical Patients With Anterior Knee Pain
Brief Title: Spring Loaded Tri-Compartment Unloader Knee Brace Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Spring Loaded Tech (Unknown)
Responsible Party: Principal Investigator, Seth Sherman, Associate Professor of Orthopaedic Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62059
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-11

CONDITIONS: Anterior Knee Pain
Keywords: Knee Brace Effectiveness

STUDY DESIGN:
Intervention Model Description: Two groups. One brace (intervention) group and one no brace (control) group.
Masking Description: No one will be masked/blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No Brace Group (No Intervention): 50% of the participants in the study that will not be receiving a TCU brace.
- Tri-Compartment Unloader Brace Group (Experimental): 50% of the participants in the study that will be receiving a TCU brace.
  Interventions: Device: Tri-Compartment Unloader Brace

INTERVENTIONS:
Device: Tri-Compartment Unloader Brace — Knee brace that is designed to reduce compressive forces on all three compartments of the knee.
  Other Names: TCU Brace
  Arms: Tri-Compartment Unloader Brace Group

SUMMARY:
This study will examine clinical outcomes related to pain and function in patients with anterior knee pain (i.e. focal patella and/or trochlea cartilage defect(s), patellofemoral arthritis) before and after standard of care, non-surgical management with and without the addition of a Tri-Compartment Unloader (TCU) knee brace during activities of daily living. Randomly selected participants will wear a TCU brace for several weeks during physical therapy and activities of daily living that is designed to reduce compressive forces in all three compartments of the knee during weight-bearing flexion. Our hypothesis is that TCU bracing will improve clinical outcomes related to pain and function.

DETAILED DESCRIPTION:
Patients in this study have been identified as good candidates by their physicians. As the study procedures closely follow the standard of care procedures in place, study participation presents little additional risk above and beyond the standard of care procedures. The study was designed to present the least risk possible consistent with sound research design.

Participants in this study will undergo standard of care X-rays that will help in eligibility determination. Participants will be randomized to either group, and will have a 50% chance of receiving the brace. Outcomes will be measured at baseline (before any intervention), 6 weeks after commencing rehabilitation at Stanford, and 3 months after commencing rehabilitation at Stanford.

These outcome measures are collected using PatientiQ which is is being used at the clinic as part of standard of care. Spring Loaded Tech is providing the TCU braces for the patients in this study at no cost.

ELIGIBILITY:
Inclusion Criteria:

1. Anterior knee pain that worsens when the knee is flexed and bearing weight
2. Patellofemoral chondral defect(s) or patellofemoral arthritis detected with standard of care x-ray and/or MRI
3. Kellgren and Lawrence grade 0-3 of PF joint
4. Able to wear the TCU knee brace for a minimum of 3 hours per day
5. Over 18 years old, can understand written English
6. Coronal knee alignment within 7 degrees of neutral
7. Must be able to fit within an off-the-shelf knee brace size provided by Company
8. Must complete physical therapy through Stanford

Exclusion Criteria:

1. Surgical intervention definitely indicated (major mechanical symptoms/failed substantial previous conservative measures) on the affected knee within the next year
2. Use of another brace designed to unload the knee or manage knee pain during the study
3. Varus/Valgus joint alignment > 7 degrees
4. Inability to be fit properly in an off-the-shelf brace provided by the Company
5. BMI >40
6. Bilateral knee symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth L Sherman, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Redwood City Outpatient Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants signed informed consent, and 14 were randomized
Groups:
- Experimental: TCU Bracing: Participants will be instructed to wear a tricompartment offloader (TCU) knee brace (Levitation 2) for a minimum of 3 hours per day during activities of daily living and undergo standard of care rehabilitation protocol.
- Control: Participants will undergo standard of care rehabilitation protocol only.
Period: Overall Study
Arm/Group | Experimental: TCU Bracing | Control
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: TCU Bracing: Participants will be instructed to wear a TCU knee brace (Levitation 2) for a minimum of 3 hours per day during activities of daily living and undergo standard of care rehabilitation protocol.
- Total: Total of all reporting groups
Arm/Group | Experimental: TCU Bracing | Control | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS) patient-reported outcome questionnaire; responses are scaled to a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Time Frame: Baseline, 6-weeks, and 3-months
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: TCU bracing | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline: number analyzed (Participants) | 2 | 5
  Baseline | 61.91 (14.42) | 72.59 (15.72)
  6 weeks: number analyzed (Participants) | 6 | 4
  6 weeks | 71.17 (8.87) | 85.99 (16.60)
  3 months: number analyzed (Participants) | 5 | 4
  3 months | 72.39 (11.19) | 86.76 (13.39)

2. Primary Outcome: Pain Visual Analog Scale (VAS)
Description: Visual Analog Scale (VAS) is rated on a scale of 0 to 100 where 0 means no pain and 100 means severe pain.
Time Frame: Baseline, 6-weeks, and 3-months
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: TCU bracing | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline: number analyzed (Participants) | 1 | 4
  Baseline | 20 (0) | 36.17 (23.37)
  6 weeks: number analyzed (Participants) | 6 | 4
  6 weeks | 12.61 (7.52) | 8.42 (10.48)
  3 months: number analyzed (Participants) | 5 | 4
  3 months | 12.33 (9.71) | 15.5 (17.92)

3. Secondary Outcome: Quality of Life (EQ-5D)
Description: Quality of life (EQ-5D) has 5 response levels where level 1 equates to no problems and level 5 equates to severe problems. The EQ-5D assesses quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses are then scaled to a score of 0 to 100 (high scores correspond to higher health related quality of life).
Time Frame: Baseline, 6-weeks, and 3-months
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: TCU bracing | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline: number analyzed (Participants) | 2 | 4
  Baseline | 67.5 (3.54) | 79.8 (12.76)
  6 Weeks: number analyzed (Participants) | 6 | 4
  6 Weeks | 74.83 (14.32) | 71.0 (32.99)
  3 Months: number analyzed (Participants) | 5 | 4
  3 Months | 85.8 (12.89) | 69.0 (26.80)

4. Secondary Outcome: Lower Extremity Activity Scale (LEAS)
Description: Lower Extremity Activity Scale (LEAS) measures daily physical activity by having patients answer 20 questions, choosing from 18 options of activity levels (0 = no activity, to 18 = college/professional athlete level of activity). Individual scores are summed and averaged to create the overall score (range: 0 to 18, with highest scores corresponding to highest level of activity).
Time Frame: Baseline, 6-weeks, and 3-months
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: TCU bracing | Control
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline: number analyzed (Participants) | 2 | 3
  Baseline | 9 (5.66) | 12.3 (5.7)
  6 Weeks: number analyzed (Participants) | 6 | 4
  6 Weeks | 13 (4.2) | 12 (4.5)
  3 Months: number analyzed (Participants) | 5 | 4
  3 Months | 14 (3.54) | 11.25 (4.57)

5. Secondary Outcome: Quadricep Strength (Girth)
Description: Using a biodex to measure quad strength.
Time Frame: Baseline; 6-weeks and 3-months post-intervention
Reporting Status: Not Posted

6. Secondary Outcome: Effusion Grade
Description: Checking how much fluid is around the knee. There are different grades. Grade 1 means no fluid-wave while performing a downward stroke whereas Grade 5 means excess of fluid that makes it impossible to stroke the medial fluid away.
Time Frame: Baseline; 6-weeks and 3-months post-intervention
Reporting Status: Not Posted

7. Secondary Outcome: Painful Crepitus With Deep Knee Flexion
Description: Painful crepitus is when there is a sensation or noise when you move a joint.
Time Frame: Baseline; 6-weeks and 3-months post-intervention
Reporting Status: Not Posted

8. Secondary Outcome: Knee Range of Motion
Description: Knee range of motion is measured at 0º extension (completely straight leg) to 130º, a fully flexed leg.
Time Frame: Baseline; 6-weeks and 3-months post-intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Experimental: TCU Bracing | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT05428332/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT05428332/SAP_001.pdf